CLINICAL TRIAL: NCT06958159
Title: Hybrid Endoscopic Stricturotomy Plus Balloon Dilation Versus Endoscopic Stricturotomy Alone for Short Strictures (<3 cm) in Crohn's Disease (The HEIST Study)
Brief Title: Hybrid Endoscopic Stricturotomy Plus Balloon Dilation Versus Stricturotomy Alone for Short Crohn's Disease Strictures
Acronym: HEIST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIG/IEC-BH&R 65/12.2024-04
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-04

CONDITIONS: Crohn Disease (CD)
Keywords: Endoscopic balloon dilation; Endoscopic stricturotomy; Crohn disease; re-intervention
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In this study, the outcomes assessors are blinded to group allocation. The individuals responsible for evaluating clinical outcomes-such as symptom recurrence, need for reintervention, hospitalization, emergency department visits, and surgical referral-are not involved in the endoscopic procedures and are unaware of which treatment (stricturotomy alone vs. hybrid therapy) the participant received. This masking is maintained throughout data collection and analysis to minimize bias in the assessment of primary and secondary outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic Stricturotomy Alone (Experimental): Participants in this arm will undergo endoscopic stricturotomy alone for the treatment of short (<3 cm), fibrotic, symptomatic Crohn's disease strictures. The procedure will be performed using a needle knife or insulated-tip knife during colonoscopy, following a standardized protocol.
  Interventions: Procedure: Endoscopic Stricturotomy
- Hybrid Endoscopic Stricturotomy Plus Balloon Dilation (Experimental): Participants in this arm will undergo hybrid therapy consisting of endoscopic stricturotomy followed by controlled radial expansion balloon dilation of the stricture during the same session. The procedure is intended to enhance luminal patency and reduce the risk of recurrence.
  Interventions: Procedure: Endoscopic Stricturotomy; Procedure: Endoscopic Balloon Dilation

INTERVENTIONS:
Procedure: Endoscopic Stricturotomy — Endoscopic stricturotomy is performed using either a needle knife or an insulated-tip (IT) knife (Olympus, Tokyo, Japan), selected based on the location and morphology of the stricture. Electrosurgical cutting is delivered using the Endo Cut I mode on an ERBE VIO 300D or VIO 3 electrosurgical unit (Erbe Elektromedizin, Germany), with standardized settings: Effect 3, Cut Duration 1, Cut Interval 3.
  Radial incisions are initially made across the stricture, followed by circumferential cutting in non-ulcerated areas to relieve luminal narrowing. The goal is to achieve adequate stricture opening while minimizing the risk of perforation.
Procedure: Endoscopic Balloon Dilation — Endoscopic balloon dilation is performed using a Controlled Radial Expansion (CRE) balloon (Boston Scientific, USA). The size of the balloon is selected based on the estimated diameter of the stricture, presence or absence of ulceration, and the anatomical location.
  The balloon is gradually inflated under endoscopic visualization to a maximum diameter of 12-20 mm, tailored to the baseline luminal narrowing. The balloon is maintained at full inflation for 60 seconds to achieve controlled and uniform dilation of the stricture.
  Arms: Hybrid Endoscopic Stricturotomy Plus Balloon Dilation

SUMMARY:
Crohn's disease is a chronic condition that can lead to inflammation and narrowing (strictures) of the intestine, causing symptoms like pain, bloating, and difficulty with bowel movements. These strictures are often treated with endoscopic procedures such as balloon dilation or stricturotomy to widen the narrowed segments and relieve symptoms.

The HEIST Study is a randomized clinical trial designed to compare two endoscopic treatment strategies for short Crohn's disease-related strictures (less than 3 centimeters in length). One group will undergo endoscopic stricturotomy alone, while the other group will receive a combination of stricturotomy followed by balloon dilation (hybrid approach).

The goal is to determine whether the hybrid approach improves long-term outcomes such as symptom relief, reduced need for repeat procedures, and avoidance of surgery. Patients will be followed for 12 months after treatment to assess durability of response, quality of life, and any complications or additional interventions needed.

This study aims to provide high-quality evidence to guide endoscopic treatment of intestinal strictures in Crohn's disease and to help identify the most effective and safest approach for long-term symptom control.

DETAILED DESCRIPTION:
The HEIST Study (Hybrid Endoscopic Stricturotomy Plus Balloon Dilation Versus Endoscopic Stricturotomy Alone for Short Strictures in Crohn's Disease) is a prospective, randomized controlled trial designed to compare two endoscopic treatment strategies for short, fibrotic strictures in patients with Crohn's disease. The trial specifically evaluates whether the addition of balloon dilation to endoscopic stricturotomy improves clinical outcomes compared to stricturotomy alone.

Eligible patients will have symptomatic, non-angulated strictures less than 3 centimeters in length, located in the colon or neo-terminal ileum. Participants will be randomly assigned during colonoscopy to receive either (1) endoscopic stricturotomy alone or (2) endoscopic stricturotomy followed by balloon dilation using a controlled radial expansion balloon (up to 18 mm diameter). Interventions will be performed using a therapeutic colonoscope and either a needle knife or insulated-tip knife, followed by balloon inflation if applicable.

All procedures will be carried out by experienced interventional endoscopists using a standardized protocol. Patients will be evaluated at baseline, immediately post-procedure, and at 1, 3, 6, and 12 months following the intervention. The follow-up includes clinical symptom scoring using the Crohn's Disease Obstructive Symptom Score, adverse event monitoring, quality of life assessment, and documentation of any further endoscopic or surgical intervention.

The primary outcome is the rate of clinical success at 12 months, defined as sustained symptom improvement without the need for repeat endoscopic or surgical intervention. Secondary outcomes include technical success, rate of complications (e.g., bleeding, perforation), time to re-intervention, and changes in quality of life metrics.

By evaluating these two commonly used endoscopic techniques in a randomized design with 12-month follow-up, the HEIST Study aims to provide evidence to optimize endoscopic treatment of short strictures in Crohn's disease and support treatment decisions in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years.
* Diagnosed Crohn's disease based on clinical, endoscopic, histologic, or radiologic criteria.
* Presence of fibrotic or mixed strictures measuring less than 3 cm in length.
* A maximum of two strictures per patient.
* Strictures located in endoscopically accessible sites

Exclusion Criteria:

* Predominantly ulcerated or active inflammatory strictures.
* Strictures longer than 3 cm.
* Strictures not accessible via standard colonoscopy.
* Pregnancy.
* Three or more strictures identified in a single patient.
* Prior endoscopic stricturotomy at the same stricture site.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Time to Clinical Recurrence Within 12 Months | Up to 12 months post-procedure
  Clinical recurrence is defined as a Crohn's Disease Obstruction Score (CDOS) >2 following an initial clinical response. Initial response is defined as a ≥2-point reduction in CDOS or normalization to CDOS ≤2. Time to recurrence is measured from the date of the procedure to the first recurrence event. Participants without recurrence will be censored at their last follow-up or at 12 months.

SECONDARY OUTCOMES:
Technical Success | Day of procedure
  Technical success is defined as the ability to pass a pediatric colonoscope beyond the treated stricture during the same session as the endoscopic procedure.
Clinical Response | 1 month post-procedure
  Clinical response is defined as a reduction in CD Obstruction Score (CDOS) by ≥2 points from baseline, or normalization of the CDOS to ≤2, measured at 1 month after the intervention.
Time to Re-intervention | Up to 12 months post-procedure
  Time (in days) from the index procedure to the first repeat endoscopic intervention (balloon dilation or stricturotomy or hybrid) for the same stricture. Participants without re-intervention will be censored at last follow-up or at 12 months
Time to Intestinal Surgery | Up to 12 months post-procedure
  Time from the index endoscopic procedure to intestinal surgery related to the treated stricture. Participants who do not undergo surgery will be censored at the last follow-up or 12 months.
Time to Stricture-Related Hospitalization | Up to 12 months post-procedure
  Time from the index procedure to first hospitalization caused by stricture-related complications or obstructive symptoms. Participants without hospitalization will be censored at last follow-up or 12 months.
Time to Stricture-Related Emergency Department Visit | Up to 12 months post-procedure
  Time from the index endoscopic procedure to the first emergency department visit related to stricture-associated symptoms. Participants without an emergency visit will be censored at last follow-up or 12 months.
Adverse events | Up to 30 days post-procedure
  Number and type of adverse events (e.g., bleeding, perforation, post-procedure pain, infection) occurring during or within 30 days of the endoscopic procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Asian Institute of Gastroenterology, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this is a single-center, investigator-initiated trial without a formal data-sharing infrastructure. De-identification and secure long-term storage mechanisms are not currently available for external data distribution. Summary-level data will be published in peer-reviewed journals.

REFERENCES:
- [Background] Lan N, Shen B. Endoscopic Stricturotomy Versus Balloon Dilation in the Treatment of Anastomotic Strictures in Crohn's Disease. Inflamm Bowel Dis. 2018 Mar 19;24(4):897-907. doi: 10.1093/ibd/izx085. PMID 29546384